CLINICAL TRIAL: NCT02147912
Title: Evaluation of Depression In Chronic Obstructive Pulmonary Disease: a Longitudinal Randomized Controlled Trial.
Brief Title: Evaluation of Depression In Chronic Obstructive Pulmonary Disease
Acronym: EDIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Catania (Other)
Responsible Party: Principal Investigator, Prof. Eugenio Aguglia, Full Professor of Psychiatry, University Hospital, Catania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHCatania
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Depression in Patients With Chronic Obstructive Pulmonary Disease
Keywords: Depression; COPD; Aerobic Exercise; Anxiety; Quality of life; neurocognitive functioning
MeSH Terms: conditions — Depression; Pulmonary Disease, Chronic Obstructive; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic exercise (Active Comparator): A six week aerobic exercise intervention in COPD depressed population.
  Interventions: Other: Aerobic Exercise
- Control sample (No Intervention): Only participants randomized in the arm named "Aerobic exercise" will receive a six weeks aerobic exercise intervention.

INTERVENTIONS:
Other: Aerobic Exercise — Aerobic exercise intervention consists of lower (treadmill and cyclette) and upper arts (arm ergometer Davenbike®) training, as well as calisthenic exercises with increasing intensity from a minimum of 80% to a maximum workload for lower arts in a minimum time.
  Arms: Aerobic exercise

SUMMARY:
Background:

Several clinical studies show high rates of anxiety and depressive disorders in Chronic Obstructive Pulmonary Disease (COPD), that suggest common underlying pathogenetic mechanisms of COPD and depressive disorders. The aim of this study is to evaluate the effects of aerobic exercise, proposed in the context of pulmonary rehabilitation, in a sample of COPD depressed patients without psychopharmacological treatment, through the correlation of some psychopathological variables and physical/pneumological parameters.

Methods:

The investigators have designed an observational longitudinal trial. The trial will be prospective 6-weeks randomized clinical study to evaluate the impact of aerobic exercise on depressive symptoms in 154 patient affected by COPD and depression, assessed by Hamilton Depression Rating Scale (HDRS). The investigators will also monitor anxiety, quality of life and neurocognitive function.

Outcome measures:

The investigators compare the variation of HDRS total score, as primary outcome measure, in two groups (A, B) of COPD depressed patients matched for: COPD status; depressive status; age; gender. Only the participants randomized in study group A will receive a 6-weeks aerobic exercise intervention.

Statistical analysis:

All tests are two-tailed and a p value 0.05 was considered significant. The difference between the two groups will be evaluated with Student's T test for normally distributed data, and with Mann-Whitney's U test, for those with not normal distribution. The normality of distribution will be evaluated with the Kolmogorov-Smirnov test. Any correlations among the variables under evaluation will be assessed by Spearman r correlation. Variables will be compared using the Chi-squared test or Fisher exact test for categorical variables.

Discussion:

There is a strong correlation between physical activity and mental health. Several data have suggested that aerobic exercise shows significant effects, comparable to pharmacotherapy and to psychotherapy, on reducing depressive symptomatology. The goal of our study is to propose an effective intervention to reduce the risk of severe depression in this special population, evaluating the variation of HDRS total score after the aerobic exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of COPD and depression, eligibility to perform pulmonary rehabilitation according to ATS and ERS guidelines.

Exclusion Criteria:

indication to restoring treatment of airway patency and current psychopharmacological treatment (including sleeping-pills).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
variation of HDRS total score | 6 weeks after intervention phase
  we compare the variation of HDRS total score, as primary outcome measure, in two groups (A, B) of COPD depressed patients matched for: COPD status; depressive status; age; gender. Only the participants randomized in study group A will receive a 6-weeks aerobic exercise intervention.

SECONDARY OUTCOMES:
daily functioning assessment | 6 weeks after intervention phase
  Evaluation of potential benefits on: anxiety symptoms, cognitive features, daily physical function (related to physical performances and/or to psychopathological dimensions) and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Aguglia, Prof., Principal Investigator — UOPI of psychiatry - Department of clinical and molecular biomedicine - AOU Policlinico-Vittorio Emanuele. Via S. Sofia, 78 - 95124 Catania, Italy; Giuseppe Minutolo, MD, PhD, Principal Investigator — UOPI of psychiatry - Department of clinical and molecular biomedicine - AOU Policlinico-Vittorio Emanuele. Via S. Sofia, 78 - 95124 Catania, Italy; Giuseppe Catalfo, MD, Principal Investigator — UOPI of psychiatry - Department of clinical and molecular biomedicine - AOU Policlinico-Vittorio Emanuele. Via S. Sofia, 78 - 95124 Catania, Italy; Francesca Magnano S. Lio, MD, Principal Investigator — UOPI of psychiatry - Department of clinical and molecular biomedicine - AOU Policlinico-Vittorio Emanuele. Via S. Sofia, 78 - 95124 Catania, Italy; Nunzio Crimi, Prof., Principal Investigator — Pulmonary Rehabilitation Clinic - Department of clinical and molecular biomedicine - AOU Policlinico-Vittorio Emanuele. Via S. Sofia, 78 - 95124 Catania, Italy